CLINICAL TRIAL: NCT06432036
Title: RENEGADE: Radioembolization for Early Stage Renal Cell Carcinoma: An Open-Label, Prospective, Multi-Center, Phase 1/2 Safety Trial
Brief Title: Yttrium-90 (Y90) Radioembolization for the Treatment of Early Stage Renal Cell Carcinoma, The RENEGADE Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-001261; NCI-2024-03516 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-05-10; First posted 2024-05-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stage I Renal Cell Cancer; Stage II Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Specimen Handling; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (radioembolization, TheraSphere) (Experimental): Patients undergo radioembolization with TheraSphere given intra-arterially. Patients undergo angiogram during screening, SPECT scan on study and CT scan and blood sample collection throughout the study.
  Interventions: Procedure: Angiogram; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Radioembolization; Procedure: Single Photon Emission Computed Tomography; Other: Survey Administration; Radiation: Yttrium Y 90 Glass Microspheres

INTERVENTIONS:
Procedure: Angiogram — Undergo angiogram
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Radiation: Radioembolization — Undergo radioembolization
  Other Names: intra-arterial brachytherapy
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Other: Survey Administration — Ancillary study
Radiation: Yttrium Y 90 Glass Microspheres — Given intra-arterially
  Other Names: TheraSphere; Y-90 Therasphere

SUMMARY:
This phase I/II trial tests the safety, side effects and effectiveness of radioembolization with yttrium-90 (Y-90) in patients with early stage renal cell carcinoma. Y-90 is a radioactive chemical that is incorporated into millions of very tiny glass spheres. These spheres are injected into the artery that feeds the cancer. This process is called radioembolization. Y-90 radioembolization may be a safe and effective treatment for patients with early stage renal cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety and toxicity of Yttrium-90 radioembolization for renal cell carcinoma (RCC).

SECONDARY OBJECTIVES:

I. To assess tumor response and duration of response, based on Choi, Response Evaluation Criteria in Solid Tumors (RECIST), and modified RECIST criteria.

II. To assess time to disease progression. III. To assess progression free survival and overall survival. IV. To assess stability of renal function via glomerular filtration rate (GFR) and cystatin-C.

V. To describe the difference in quality of life before and after treatment using Eastern Cooperative Oncology Group (ECOG) performance status and RCC-specific Quality of Life (QoL) questionnaire.

OUTLINE:

Patients undergo radioembolization with yttrium Y 90 glass microspheres (TheraSphere) given intra-arterially. Patients undergo angiogram during screening, single proton emission computed tomography (SPECT) scan on study and computed tomography (CT) scan and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 1 day, 1 week, and then monthly for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged ≥ 18 years at the time of screening
* Written informed consent and any locally required authorization (e.g., Health Insurance Portability and accountability Act) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Life expectancy ≥ 12 months
* RCC, diagnosed by radiographic imaging and histology
* Clinical stage of RCC: T1 or T2a, Cancer stage (N0M0)
* 1-2 solid (> 80% solid) target lesions
* Patient not an ideal candidate for partial nephrectomy or thermal ablation at the time of study entry, based on the decision of the institution's multidisciplinary tumor board. Contraindications for partial nephrectomy include inability to potentially partially resect the kidney, high risk of adverse events due to medical comorbidities, or potential high risk of adverse events due to general anesthesia. Contraindications to thermal ablation include potential inability to technically place ablation probes into the tumor, central tumors which risk thermal injury to the renal collecting system
* Patient not considered a candidate for long-term active surveillance due to oncologic risk due to tumor growth and/or tumor size
* Patient not considered ideal candidates for radical nephrectomy due to surgical comorbidity and/or development of adverse health outcomes
* Measurable tumor by RECIST 1.1 criteria
* Absence of bilateral renal tumors
* Negative serum pregnancy test in females of child-bearing potential; patients who are breast-feeding cannot participate in this trial
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Absolute lymphocyte count ≥ 1.0 x 10^9/L
* Platelet count ≥ 75 x 10^9/L
* Glomerular filtration rate (GFR) ≥ 45 mL/min/1.73 m^2
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* Screening mapping angiogram demonstrates successful localization of tumor(s), where catheter placement location(s) would allow Y90 to distribute in the intended treatment area, without venous shunting

Exclusion Criteria:

* Any contraindication to angiography or selective renal artery catheterization
* Screening angiography with cone beam CT (CBCT) shows any arterial flow to the gastrointestinal tract uncorrectable by angiographic techniques
* Screening angiography with CBCT shows poor tumor targeting that would lead to a dose that does not meet the renal dosing criteria. This typically occurs when a feeding artery to the tumor cannot be identified
* Screening angiography demonstrates excessive non-tumoral renal parenchyma will be in the treatment field, that the new baseline glomerular filtration rate will be < 45 mL/min/1.73 m^2
* Screening angiography demonstrates renal venous shunting of iodinated contrast that is immediately visible upon arterial injection
* Extra-renal metastases, including patients with abdominal lymph nodes >1.5 cm in shorter axis, or with lung nodules (single lesion, >1 cm, or multiple smaller lesions with a total diameter >2 cm)
* Brain metastases, leptomeningeal carcinomatosis or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
* Evidence of any tumor invasion into the renal vein, renal artery, or renal collecting system
* Any prior radiation therapy to the abdomen, including localized radiation therapy to the index tumor
* Concurrent treatment for RCC or treatment in the last 6 months in another clinical study, unless it is an observational study (non-interventional) or during a non-interventional follow-up stage of an interventional study, or prior randomization to this study
* History of active primary/acquired immunodeficiency
* Presence of renal ureteral stent in the treatment kidney at any time
* History of malignancy, other than RCC, within three years, with the exception of adequately treatment carcinoma in situ of the cervix, early squamous cell carcinoma or basal cell carcinoma of the skin, localized prostate cancer, ductal carcinoma in situ, or low-grade endometrial carcinoma with no myometrial invasion (negligible risk of metastases or death 5-year overall survival [OS] rate > 90%)
* Major surgical procedure (as defined by the Investigator) within 28 days prior to enrollment
* A history of severe allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically
* Active infection
* Female patients who are pregnant or breastfeeding or female patients of reproductive potential who are not willing to employ effective birth control from screening to 6 months after treatment
* Unstable chronic disease or evidence of any disease or condition that would place the patient at undue risk and preclude safe use of Y90 microspheres, including but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* History of pulmonary insufficiency, measured by oxygen saturation of less than 90%
* Solitary kidney
* Patient not able to follow the study protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of treatment related adverse events | Up to 2 years
Number of serious adverse events | Up to 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  According to Choi, Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, and modified RECIST. Will be summarized as count and percentage. The corresponding 95% confidence interval (CI) for the ORR will be computed using the methodology of Clopper-Pearson.
Duration of response | From the first response and first observation of progressive disease, up to 2 years
  According to Choi, RECIST 1.1, and modified RECIST. Will be analyzed by Kaplan Meier methodology.
Renal time to progression | Up to 2 years
  According to Choi, RECIST 1.1, and modified RECIST. Kaplan Meier curves will be presented.
Progression free-survival | Up to 2 years
  According to Choi, RECIST 1.1, and modified RECIST. Kaplan Meier curves will be presented.
Overall survival | Up to 2 years
  Kaplan Meier curves will be presented.
Change in renal function | Up to 2 years
  Measured by glomerular filtration rate (GFR), creatinine, and cystatin-C.
Proportion of patients receiving subsequent treatment for RCC after study treatment | Up to 2 years
  Will be summarized as counts and percentage. The corresponding 95% CIs will be computed using Clopper-Pearson.
Type of subsequent RCC treatment received after study treatment | Up to 2 years
  Will be summarized using descriptive summaries.
Proportion of patients to undergo curative therapy | Up to 2 years
  Will be summarized as counts and percentage. The corresponding 95% CIs will be computed using Clopper-Pearson.
Time to subsequent RCC treatment (local or systemic therapy) | Up to 2 years
  Will be summarized using descriptive summaries.
Correlation between tumoral absorbed dose, with efficacy and safety | Up to 2 years
  Correlation between tumoral absorbed dose (measured in Gy based on SPECT-CT) and safety (measured by incidence of Grade 3/4 treatment-related adverse events) and efficacy (measured by partial and complete response using Choi/mRECIST/RECIST criteria on follow up cross sectional imaging)
Correlation between normal tissue absorbed dose, with efficacy and safety | Up to 2 years
  Correlation between normal tissue absorbed dose (measured in Gy based on SPECT-CT) and safety (measured by incidence of Grade 3/4 treatment-related adverse events) and efficacy (measured by partial and complete response using Choi/mRECIST/RECIST criteria on follow up cross sectional imaging)
Change in Eastern Cooperative Oncology Group score | Up to 2 years
  The scale is Eastern Cooperative Oncology Group (ECOG). Scale is 1 to 5, with 5 being the worst outcome.
Change in quality of life as measured by the SF-36 (QualityMetrics) Quality of Life survey | Up to 2 years
  Change in overall quality of life based on patient-reported outcomes
Percentage of subjects with absorbed Y90 dose within range (+/- 20%) of planned dose | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth A Padia, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Meiselman S, Thomas MA, Giardina JD, Zheleznyak A, Thorek DLJ, Malone CD. Advances in Radioembolization for Liver Cancer. J Vasc Interv Radiol. 2025 Dec;36(12):1876-1881. doi: 10.1016/j.jvir.2025.07.018. PMID 41276366